CLINICAL TRIAL: NCT07254208
Title: A Long-term Observational Study in Participants Who Have Received PBGENE-HBV, an In Vivo Gene Editing Investigational Product, in a Prior Clinical Study
Brief Title: A Long-term Observational Study in Participants Who Have Received PBGENE-HBV
Acronym: ELIMINATE-B
Status: Not yet recruiting | Type: Observational
Sponsor: Precision BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PBGENE-HBV-02
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Chronic HBV Infection
Keywords: Hepatitis B Chronic; Gene Therapy; Gene Editing; PBGENE-HBV
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: PBGENE-HBV — PBGENE-HBV is the investigational product administered in the parent study. This LTFU study is non-interventional; no investigational product given.

SUMMARY:
Participants who received at least one dose of PBGENE-HBV will be enrolled in this LTFU study.

DETAILED DESCRIPTION:
This is a LTFU observational study designed to evaluate the safety of PBGENE-HBV in participants previously exposed to PBGENE-HBV. This study protocol does not include administration of PBGENE-HBV.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has received at least 1 dose of PBGENE-HBV investigational product in a prior clinical study
2. Participant, or their legally authorized representative, has provided signed informed consent.

Exclusion Criteria:

* N/A

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received at least one dose of PBGENE-HBV will be enrolled in this LTFU study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2040-01 (Estimated); Study Completion 2040-06 (Estimated)

PRIMARY OUTCOMES:
Safety to assess frequency, severity, and outcome of delayed adverse events | 15 years
  Delayed adverse events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Interventional Study PBGENE-HBV-01 — https://clinicaltrials.gov/study/NCT06680232?term=NCT06680232&rank=1